CLINICAL TRIAL: NCT04193566
Title: Acute Effects of Sodium-glucose Cotransporter-2 Inhibition on Renal Oxygenation and Autonomic Function in Type 1 Diabetes
Brief Title: Acute Effects of SGLT2 Inhibition on Renal Oxygenation and Autonomic Function in Type 1 Diabetes
Acronym: Astronaut
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-19052662; 2019-004557-92 (EudraCT Number)
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Nephropathy; Hypoxia; Mitochondrial Alteration; Type 1 Diabetes; Autonomic Neuropathy, Diabetic
MeSH Terms: conditions — Kidney Diseases; Hypoxia; Diabetes Mellitus, Type 1; Diabetic Neuropathies | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, placebo-controlled, cross-over intervention study
Who Masked: Participant, Investigator
Masking Description: Group allocation is concealed to patients as well as investigators. 60 sequentially numbered, opaque, sealed envelopes will be produced by Glostrup Apotek. All persons involved in the conduct of the study are blinded to the randomization code. Randomization codes and envelopes are stored securely at the study site available only for the unblinded site staff in charge of randomizing subjects and dispensing study products to subjects. Sealed codes are marked according to randomization code and distributed according to a pre-distributed order. Should unblinding of a study participant be necessary because of an emergency, a dedicated person at Steno Diabetes Center Copenhagen, not involved in the study, will perform the procedure. Alternatively, the Principal investigator will be able to perform unblinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): Patients in the active arm will be treated with dapagliflozin 50 mg once on site for visit 2 and once at home on the evening before visit 3.
  Forxiga®, dapagliflozin 10 mg film-coated tablet.
  For further information please refer to:
  https://www.ema.europa.eu/en/documents/product-information/forxiga-epar-product-information_en.pdf.
  Interventions: Drug: Forxiga
- Placebo (Placebo Comparator): Patients in the placebo arm will be treated with placebo once on site for visit 2 and once at home on the evening before visit 3.
  Placebo drug:
  The composition equals the composition of Forxiga® - just with the active ingredient omitted. Active drug and placebo are similar in appearance and smell.
  Interventions: Drug: Forxiga

INTERVENTIONS:
Drug: Forxiga — Forxiga®, dapagliflozin 10 mg film-coated tablet.
  For further information please refer to:
  https://www.ema.europa.eu/en/documents/product-information/forxiga-epar-product-information_en.pdf.
  Common side effects include hypoglycemia, hypotension, elevated hematocrite, dyslipidemia, back pain, dizziness, skin rash, urinary tract infection, vulvovaginitis and dehydration. Very rare incidents of ketoacidosis have been observed. Side effects have only been observed after use in longer periods and not in single-dose usage, as planned in the present study. A dose of 50 mg has been chosen to achieve optimal efficacy. Once-per-day doses of dapagliflozin for 12 weeks of 2.5 mg, 5 mg, 10 mg, 20 mg and 50 mg have been demonstrated to be relatively safe across the mentioned doses (20) and no apparent risk is expected from instituting two single-doses of 50 mg dapagliflozin.
  Other Names: dapagliflozin

SUMMARY:
Background: Inhibiting the sodium-glucose cotransporter-2 (SGLT2) has been observed to reduce risk of cardiovascular events and kidney failure in type 2 diabetes. The exact mechanisms of the beneficial effects of SGLT2 inhibition (SGLT2i) are still unknown. Kidney hypoxia has been demonstrated in diabetic kidney disease and SGLT2i is thought to relieve hypoxia in the kidneys. Mitochondrial dysfunction and autonomic dysfunction might also contribute to kidney hypoxia.

Objective: The primary aim of the study is to assess the acute effects of SGLT2 inhibition on parameters reflecting oxygenation and oxygen consumption of the human kidney in persons with type 1 diabetes. Exploratory aims are to investigate acute changes in oxygen availability and oxygen access to the kidneys after SGLT2i. This include measures of peripheral blood oxygenation, mitochondrial function and autonomic function.

Methods: Acute intervention study with oral dapagliflozin given in two doses each of 50 mg or matching placebo as intervention. Kidney oxygenation and perfusion parameters will be assessed by blood-oxygen-dependant level magnetic resonance imaging. Mitochondrial function will be assessed by extracellular flux analysis on lymphocytes. Autonomic function will be assessed by measuring baroreflex sensitivity.

Design: Randomized, double blinded, placebo-controlled, cross-over intervention study.

Study population: Fifteen healthy controls are recruited by advertisement and 15 patients with type 1 diabetes recruited from Steno Diabetes Center Copenhagen.

Endpoints: Primary end-point: Renal cortical and medullary oxygenation (T2*). Exploratory end-points: Renal cortical and medullary perfusion, renal artery flow, renal oxygen consumption, peripheral capillary oxygen saturation (SpO2), arterial oxygen partial pressure (PaO2), arterial oxygen saturation (SaO2), lymphocyte mitochondrial function, baroreflex sensitivity.

Timeframe: Inclusion of patients from January 2020. Last patient last visit January 2021. Data analysis completed spring 2021, presentation autumn 2021 and publications Winter 2021.

ELIGIBILITY:
Inclusion criteria healthy controls:

* Written informed consent must be provided before participation
* Male or female patients > 18 years of age
* Capable of lying in a MR-scanner for two hours

Inclusion criteria persons with type 1 diabetes:

* Written informed consent must be provided before participation
* Male or female patients >18 years of age with a diagnosis of type 1 diabetes (WHO criteria)
* Urinary albumin creatinine ratio (UACR) ≥30 mg/g in 2 out of 3 consecutive samples (albuminuria) prior to randomization assessed from electronic laboratory database.
* Capable of lying in a MR-scanner for two hours

Exclusion criteria for all:

* Non-diabetic kidney disease as indicated by medical history and/or laboratory findings
* Renal failure (eGFR<15 ml/min/1.73m2), dialysis or kidney transplantation
* Treatment with beta-blocking medication
* Uncontrolled arrhythmia, 2. or 3. degree AV-block or sick sinus syndrome - assessed from a standard 12-lead electrocardiogram
* Pregnancy or breastfeeding (urine HCG is performed on all fertile women)
* Systolic blood pressure < 90 or > 200 mmHg
* Patients who, in the judgement of the investigator, is incapable of participating
* Exclusion criteria for MRI

  * Claustrophobia
  * Known heart disease
  * Known lung disease
  * Have had surgery the past six weeks
  * Have foreign bodies of metal in the body (e.g. pacemaker, metal plates, metal screws)
* Exclusion criteria for arterial blood gas sampling (only patients with type 1 diabetes)

  * Absent pulse
  * Raynauds syndrome
  * Buergers Disease (thromboangiitis obliterans)
  * Inadequate or interrupted circulation
  * Anticoagulation treatment
  * Coagulopathies (hypo or hyper coagulable states)
  * Arterial atherosclerosis
  * Insufficient collateral perfusion
  * Partial or full thickness burns over the cannulation site
  * Synthetic arterial or vascular grafts or infection at the proposed site of cannulation Patients with type 1 diabetes will have the possibility to participate in the study without getting arterial blood gas sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Renal oxygenation | From baseline to +3 hours from intervention
  Blood Oxygen Level Dependent (BOLD) Magnetic Resonance Imaging (MRI) assessing the transverse relaxation time of atomic nuclei in the tissue (T2*) in miliseconds (ms).
Change in Renal oxygenation | From baseline to +6 hours from intervention
  BOLD MRI assessing the transverse relaxation time of atomic nuclei in the tissue (T2*) in miliseconds (ms).

SECONDARY OUTCOMES:
Change in renal cortical and medullary perfusion | From baseline to +3 hours from intervention
  Renal tissue perfusion can be measured noninvasively with MRI using arterial spin labelling (ASL). It is measured in mL/g/min.
Change in renal cortical and medullary perfusion | From baseline to +6 hours from intervention
  Renal tissue perfusion can be measured with MRI using arterial spin labelling (ASL). It is measured in mL/g/min.
Change in renal artery flow | From baseline to +3 hours from intervention
  Renal artery flow can be measured by using phase contrast (PC) MRI. It is measured in mL/min.
Change in renal artery flow | From baseline to +6 hours from intervention
  Renal artery flow can be measured by using phase contrast (PC) MRI. It is measured in mL/min.
Change in renal oxygen consumption | From baseline to +3 hours from intervention
  Renal oxygen consumption can be measured using Q-flow combined with BOLD MRI. It is measured in pmol/min/microgram protein.
Change in renal oxygen consumption | From baseline to +6 hours from intervention
  Renal oxygen consumption can be measured using Q-flow combined with BOLD MRI. pmol/min/microgram protein
Change in peripheral capillary oxygen saturation (SpO2) | From baseline to +3 hours from intervention
  Pulse oximetry on index finger of the right hand. Estimates blood oxygen saturation from capillary blood. Measured in %.
Change in peripheral capillary oxygen saturation (SpO2) | From baseline to +6 hours from intervention
  Pulse oximetry on index finger of the right hand. Estimates blood oxygen saturation from capillary blood. Measured in %.
Change in blood oxygen partial pressure (PaO2) | From baseline to +3 hours from intervention
  Blood gas analysis on arterial blood. Measured in kPa.
Change in blood oxygen partial pressure (PaO2) | From baseline to +6 hours from intervention
  Blood gas analysis on arterial blood. Measured in kPa.
Change in arterial blood oxygen saturation | From baseline to +3 hours from intervention
  Blood gas analysis on arterial blood. Measured in %.
Change in arterial blood oxygen saturation | From baseline to +6 hours from intervention
  Blood gas analysis on arterial blood. Measured in %.
Change in Peripheral Blood Monocyte mitochondrial function | From baseline to +12 hours from intervention
  Seahorse X96 analyzer. Analyzes the oxygen consumption rate (OCR), measured in pMoles/min.
Change in levels of circulating inflammatory markers | From baseline to +12 hours from intervention
  Commercially available panel from the company Olink. Includes 92 biomarkers. Information on the panel can be found here: https://www.olink.com/products/inflammation/#.
Change in baroreflex sensitivity | From baseline to +12 hours from intervention
  Calculated from continous blood pressure and the distance between the R-waves in a continuous ecg. Baroreflex sensitivity describes how much heart-rate changes when blood pressure changes. Assessment of baroreflex sensitivity is done in a measurement of 5 minutes. The unit is ms/mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laursen JC, Sondergaard-Heinrich N, de Melo JML, Haddock B, Rasmussen IKB, Safavimanesh F, Hansen CS, Storling J, Larsson HBW, Groop PH, Frimodt-Moller M, Andersen UB, Rossing P. Acute effects of dapagliflozin on renal oxygenation and perfusion in type 1 diabetes with albuminuria: A randomised, double-blind, placebo-controlled crossover trial. EClinicalMedicine. 2021 Jun 28;37:100895. doi: 10.1016/j.eclinm.2021.100895. eCollection 2021 Jul. PMID 34386735

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT04193566/Prot_SAP_000.pdf